CLINICAL TRIAL: NCT03512665
Title: Impact of a Supplement of Vegetable Oils on Body Weight and Composition, Insulin Sensitivity and Other Cardiovascular Risk Factors in People at Risk of Developing Type 2 Diabetes Mellitus.
Brief Title: Evaluation of the Impact of a Nutritional Supplement Made of Vegetable Oils in People at Risk of Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Los Andes, Columbia (Other)
Collaborators: Team Foods Colombia S.A. (Industry)
Responsible Party: Principal Investigator, Carlos O Mendivil, Associate Professor, School of Medicine, University of Los Andes, Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TFC-111-2017
Record Dates: First submitted 2018-04-18; First posted 2018-05-01 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Insulin Resistance
Keywords: Pre-diabetes; cardiovascular risk; lipids; insulin resistance; obesity; overweight
MeSH Terms: conditions — Insulin Resistance; Glucose Intolerance; Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Full dose supplement group (Experimental): Patients assigned to this group will receive a daily dose of 7 mL of the study supplement (a mixture of pine, macadamia and pomegranate oils). The appearance and organoleptic properties will be similar to those of the interventions in the other two groups
  Interventions: Dietary Supplement: Full dose supplement
- Low dose Supplement group (Experimental): Patients assigned to this group will receive a daily dose of 7 mL of a mixture containing 50% study supplement and 50% sunflower oil. The appearance and organoleptic properties will be similar to those of the interventions in the other two group
  Interventions: Dietary Supplement: Low dose Supplement
- Control Oil Group (Other): Patients assigned to this group will receive a daily 7 mL dose of an oil (sunflower oil) with appearance and organoleptic properties similar to those of the supplement provided in the intervention groups
  Interventions: Other: Control Oil

INTERVENTIONS:
Dietary Supplement: Full dose supplement — A 7ml vial composed of a mixture of pine, macadamia and pomegranate oils.
  Arms: Full dose supplement group
Dietary Supplement: Low dose Supplement — A 7 mL vial composed of a mixture containing 50% study supplement (Pine, macadamia and pomegranate oils) and 50% sunflower oil.
  Arms: Low dose Supplement group
Other: Control Oil — A 7ml vial composed of sunflower oil with appearance and organoleptic properties similar to those of the supplement provided in the intervention groups.
  Arms: Control Oil Group

SUMMARY:
Metabolic and cardiovascular diseases are the first cause of morbidity and mortality throughout the world, including Latin America and Colombia. Asymptomatic elevations of blood glucose, insufficient response to normal insulin concentrations (called insulin resistance), overweight and obesity can cause severe damage to body organs, leading to complications and even death. Worryingly, the prevalence of prediabetes is on the rise and efforts in public health policies made to contain this epidemic have had a very limited impact. This has prompted an intense search for non-pharmacological interventions. One of the most promising areas is research on "nutraceuticals", foods capable of positively impacting risk factors. However, there are insufficient nutritional or supplementary alternatives to favorably impact carbohydrate metabolism and cardiovascular risk factors in individuals at risk of diabetes. This project will evaluate the effects of the administration of a dietary supplement composed of vegetable oils. The fat composition of these oils is likely to impact positively on the metabolic profile of subjects at risk of diabetes and cardiovascular conditions.

DETAILED DESCRIPTION:
Chronic non-communicable diseases (NCDs) account for 63% of deaths worldwide, of which 80% occur in low- and middle-income countries In Colombia, 71% of all deaths are related to NCDs . This pandemic can be prevented by controlling the risk factors, seeking to create interventions that impact more than one risk factor at a time, including body weight, blood glucose levels, blood pressure, cardiorespiratory fitness and other relatively minor risk factors.

On the other hand, diabetes mellitus is a major cause of morbidity and mortality worldwide . In its natural history, diabetes is preceded by factors that confer risk of diabetes and for a group of disorders known as "prediabetes" term comprising intolerance carbohydrates and impaired fasting glycaemia . Although people at risk of diabetes or prediabetes are often asymptomatic; lesions develop in micro and macrovascular beds and result in long-term kidney dysfunction, retinal damage and affectation of peripheral nerves and arteries. Vascular damage leads to an increased risk of retinopathy renal insufficiency , painful or autonomic neuropathy and atherosclerotic cardiovascular threatening diseases such as acute myocardial infarction.

The above situation has prompted an intense search for non-pharmacological interventions to intervene in patients at risk of diabetes and prevent negative consequences on the body in the short, medium and long term. One of the most promising areas of research is the nutraceuticals field. Colombian Team Foods S.A has developed a supplement of vegetable oils, that for their composition could have the ability to improve pathophysiological phenomena associated with the development of diabetes and its complications.

The main objective of this trial is to assess the impact of the consumption of a vegetable oils-based designed jointly by Team Foods and university of los Andes, on several indicators metabolic health in people at risk of diabetes. The specific objectives are:

* To enroll a sample of patients who are at risk of diabetes but have not receive drugs to control plasma glucose, cholesterol or triglycerides, and have not developed complications like kidney or eye dysfunction.
* To evaluate the effect of daily consumption of the study supplement on fasting blood glucose, the area under the glucose curve in an oral glucose tolerance test, and glycated hemoglobin (HbA1c-an indicator of blood glucose levels over the last 3 months).
* To evaluate the effect of the supplement on indexes and biomarkers of insulin resistance.
* To evaluate the effect of the supplement on other cardiovascular risk factors including lipid profile, blood pressure, body weight and body composition.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Risk of type 2 diabetes (T2DM) given by BMI 25 kg/m2 or greater and / or Finnish Diabetes Risk Score(FinnRisc) greater than 12.
* Manifest desire to participate in the study, and provision of informed consent.
* Participants must continue their regular eating habits and physical activity.

Exclusion Criteria:

* Current participation in a systematic weight loss program.
* Current use of medications that modify insulin sensitivity (except contraceptives in the case of women).
* Known hypersensitivity to any component of the supplement.
* Gastrointestinal problems that negatively affect the adherence to the study intervention.
* Known complications from diabetes or hypertension: Coronary heart disease, nephropathy, retinopathy, cerebrovascular disease, diabetic foot or painful neuropathy.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-04-07 (Actual); Primary Completion 2018-06-16 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Homeostasis Model Assessment - Insulin Resistance (HOMA-IR) | Measured at baseline and at week 8.
  Change in the HOMA-IR index at week 8, relative to baseline. HOMA-IR is calculated as the product of the fasting glycemia in mmol/L and fasting insulinemia in microunits/mL, divided by the constant 22.5.

SECONDARY OUTCOMES:
Glycated hemoglobin A1c (HbA1c) | Measured at baseline and at week 8.
  Change in the values of HbA1c at week 8, relative to baseline
Body-mass index | Assessed at baseline and at week 8
  Change in the patients' BMI at week 8, relative to baseline
Percent body fat. | Assessed at baseline and at week 8
  Change in impedanciometry-estimated percent body fat at week 8, relative to baseline
Percent abdominal fat | Assessed at baseline and at week 8.
  Change in impedanciometry-estimated percent abdominal fat at week 8, relative to baseline.
Lean body mass. | Assessed at baseline and at week 8.
  Change in impedanciometry-estimated lean body mass.
Waist circumference. | Assessed at baseline and at week 8.
  Change in waist circumference
High-sensitivity C-reactive protein (hsCRP) | Measured at baseline and at week 8.
  Change in plasma hsCRP.
Pigment epithelium-derived factor (PEDF). | Measured at baseline and at week 8.
  Change in plasma levels of PEDF, a biomarker of insulin resistance.
Change in plasma adiponectin | Measured at baseline and at week 8
  Change in plasma levels of total adiponectin.
Change in plasma FGF-21 | Measured at baseline and at week 8.
  Change in plasma levels of Fibroblast growth factor 21 (FGF-21).

CONTACTS AND LOCATIONS:
Overall Officials: Carlos O Mendivil, MD. PhD, Principal Investigator — University of Los Andes, Columbia
Locations (1):
- University Of Los Andes Columbia, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pelaez-Jaramillo MJ, Valencia-Enciso N, Cardenas-Mojica AA, Gaete PV, Scher-Nemirovsky EA, Gomez-Arango LF, Colmenares-Araque D, Castro-Lopez CA, Betancourt-Villamizar E, Jaimes-Madrigal J, Alvarez CA, Jimenez-Mora MA, Quiroga-Padilla PJ, Puerto-Baracaldo DK, Mendivil CO. Impact of a Formulation Containing Unusual Polyunsaturated Fatty Acids, Trace Elements, Polyphenols and Plant Sterols on Insulin Resistance and Associated Disturbances. Diabetes Ther. 2020 Jan;11(1):229-245. doi: 10.1007/s13300-019-00721-z. Epub 2019 Nov 5. PMID 31691133